CLINICAL TRIAL: NCT01410461
Title: Prospective Observational Study That Evaluates Predictor Tests for the Success of Myofascial Pelvic Floor Muscles for the Treatment of PBS
Brief Title: Identifying Predictors of Treatment Success in Painful Bladder Syndrome
Acronym: PBS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Dalia Kesner, MD, Zvolon Medical Center
Other Study IDs: RMV-0232-10; RMB-0232-10 (Other: Helsinki)
Record Dates: First submitted 2011-08-04; First posted 2011-08-05 (Estimated); Last update posted 2011-08-05 (Estimated); Status verified 2011-08

CONDITIONS: Painful Bladder Syndrome
Keywords: painful bladder; physical therapy; levator ani
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with painful bladder syndrome: Patients with diagnosis of PBS Will be offered to take part in the following study.
  Interventions: Device: quantitive sensory testing; Device: Ultrasound testing

INTERVENTIONS:
Device: quantitive sensory testing — Mechanical pain threshold: Threshold will be assessed, by using the von Frey filaments. The lowest gram weight capable of inducing pain in two of three trials will be considered as a pain threshold Heat pain threshold (HPT): HPT will be measured using thermal sensory analyzer
  Other Names: TSA, Medoc Ramat Yishay, Israel
Device: Ultrasound testing — Morphological measures of the pelvic muscles: Using a 3D 4-8MHz abdominal probe ultrasound testing will be performed. The following parameters will be measured: (1) anteroposterior hiatal diameter; (2) lateral hiatal diameter; (3) levator ani thickness and length at 3 o'clock and 9 o'clock; (4) length of the obturator (5) length of the pubococcygeus muscle; (6) obturator thickness.
  Other Names: Voluson 730 Expert; GE Healthcare

SUMMARY:
Study aims to: (1) evaluate the role of morphological and physiological characteristics of the pelvic floor, pain-related psychological and -psychophysical variables in prediction of the success of myofascial physical therapy (MPT) for the treatment of painful bladder syndrome Patients with clinical symptoms of PBS will undergo physical examination, sensory testing in the genital area, perineal ultrasound examination for the evaluation of the length of the levator muscles before MPT and following 10 consecutive sessions of MPT.

Improvement in clinical symptoms will be assessed and evaluated for correlations with psychophysical examinations.

DETAILED DESCRIPTION:
Background: Chronic pelvic pain syndrome (CPPS) is highly prevalent, yet its etiology and the treatment approach are not clear. Painful bladder syndrome (PBS), a subtype of CPPS, is commonly treated by Myofascial physical therapy (MPT), however its efficiency is limited to portion of patients. The relative contribution of local factors such as pelvic anatomical and physiological function compared with systemic pain- related psychological and psychophysical parameters in the prediction of MPT outcome has not been illumined yet.

Hypothesis and aims: Assuming that MPT has mainly local effect its treatment success can be predicted by local impairment of pelvic anatomical and physiological function assessed pretreatment.

Study aims to: (1) evaluate the role of morphological and physiological characteristics of the pelvic floor, pain-related psychological and -psychophysical variables in prediction of MPT success, (2) to assess the effect of MPT on these parameters.

Methods: PBS patients will be evaluated for symptoms severity prior to MPT by: (1) pelvic physical examination for identification of trigger points, (2) self-report of pelvic pain intensity on visual analogue scale (VAS), (3) filling a questionnaire for urinary urgency symptoms, (4) evaluation of morphological and physiological characters of pelvic muscles floor by ultrasound and Doppler, respectively, (5) assessment of pain-related psychological variables (depression, somatization and pain catastrophizing) by questionnaires, and (6) psychophysical tests of experimental pain perception. Following 3 months treatment of MPT, patients will be reevaluated for the same tests. Treatment success will be determined by 30% reduction in pain and urinary urgency.

Expected results: Patients with shorter levator muscles and reduced blood flow in the pelvic region will benefit from MPT compared to patients with augmented pain sensitivity and higher depression, pain catastrophizing and somatization scores. MPT will elongate levator muscles and increased blood flow to the pelvic region that will be associated with the improvement in PBS symptoms.

Importance: The significance of the proposed study stems from its potential to extend conceptualizing of mechanisms associated with PBS and its treatment success.

ELIGIBILITY:
Inclusion Criteria:

1. age > 18 years old
2. urinary frequency of at least 10 per 24 hr including one nighttime voiding
3. complaints of bladder pain that has been present for at least 3 months
4. pain intensity rated at least four on a VAS from 0 ''no pain at all'' to 10 ''worst imaginable pain'' during the previous month
5. pelvic digital exam reveals at least three different TrPs in the levator ani muscles that are verbally confirmed.

Exclusion criteria:

1. history of pelvic cancer or radiation
2. pelvic or abdominal surgery within 3 months
3. urinary tract infection within the last month
4. diagnosis of fibromyalgia or irritable bowel disease
5. diagnosis of neurologic disorder; diabetes; pregnancy;
6. pelvic pain and/ or urgency symptoms presented only during menses.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinical diagnosis of painful bladder syndrome
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Reduction of pain level | 3 months
  Following MPT it is expected that patients PBS symptoms will be improved as will be evaluated by VAS.

SECONDARY OUTCOMES:
Elongation of levator ani muscles. | 3 months
  Following MPT treatment it is expected that the levator ani muscles will be elongated as will be measured by perineal US.

CONTACTS AND LOCATIONS:
Overall Officials: Lior Lowenstein, MD, Study Chair — Rambam Health Care Campus
Locations (1):
- Zvolon Medical Center, Haifa, Israel

REFERENCES:
- [Background] Anderson RU, Sawyer T, Wise D, Morey A, Nathanson BH. Painful myofascial trigger points and pain sites in men with chronic prostatitis/chronic pelvic pain syndrome. J Urol. 2009 Dec;182(6):2753-8. doi: 10.1016/j.juro.2009.08.033. Epub 2009 Oct 17. PMID 19837420
- [Background] FitzGerald MP, Anderson RU, Potts J, Payne CK, Peters KM, Clemens JQ, Kotarinos R, Fraser L, Cosby A, Fortman C, Neville C, Badillo S, Odabachian L, Sanfield A, O'Dougherty B, Halle-Podell R, Cen L, Chuai S, Landis JR, Mickelberg K, Barrell T, Kusek JW, Nyberg LM; Urological Pelvic Pain Collaborative Research Network. Randomized multicenter feasibility trial of myofascial physical therapy for the treatment of urological chronic pelvic pain syndromes. J Urol. 2009 Aug;182(2):570-80. doi: 10.1016/j.juro.2009.04.022. Epub 2009 Jun 17. PMID 19535099